CLINICAL TRIAL: NCT00315861
Title: A Phase I Study of Topotecan in Combination With Pemetrexed in Patients With Advanced Malignancies
Brief Title: Topotecan in Combination With Pemetrexed in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry); Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 72; 105114; H3E-US-I013 LILLY
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Lung Cancer
Keywords: ovarian carcinoma; endometrial carcinoma; cervical carcinoma; lung carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Lung Neoplasms | interventions — Pemetrexed; Topotecan

INTERVENTIONS:
Drug: pemetrexed
Drug: topotecan

SUMMARY:
Currently, no data exists regarding the safety and tolerability of a combination regimen utilizing weekly topotecan in combination with pemetrexed. Although both drugs are associated with myelosuppression, it is hoped that the utilization of the weekly topotecan dosing schedule will allow the drugs to be easily combined. This phase I trial will evaluate the safety and tolerability of weekly topotecan in combination with pemetrexed in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Three patients will be accrued at each of 5 dose levels. Dose escalation will only proceed if none of the additional 3 patients experience DLT. The highest dose level that generates DLT in 0/3 or 1/6 patients will be the maximum tolerated dose (MTD) or the doses recommended for subsequent studies. A total of 10 patients will be treated at the MTD to further assess the toxicity of the dosing regimen and its suitability for use in subsequent trials. Patients may continue to receive treatment until unacceptable toxicity or disease progression is encountered. Treatment cycles will be repeated every 21 days. The protocol is also designed to enroll an additional 10 patients at the maximum tolerated dose to increase the confidence in the safety and suitability of the doses that are chosen for subsequent studies.

* Topotecan Day 1 and 8
* Pemetrexed Day 1

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced solid tumors
* Measurable or evaluable disease
* Age ≥ 18 years
* Karnofsky performance status ≥ 80% (ECOG 0 or 1)
* Adequate liver, bone marrow and kidney function

Exclusion Criteria:

* More than 3 prior chemotherapy regimens in the metastatic setting
* Prior treatment with topotecan or pemetrexed
* Clinically significant third space fluid present at the time of treatment
* Unable to interrupt aspirin, other non-steroidal anti-inflammatory drugs
* Inability to take steroid premedications or vitamin supplementation
* The presence of active brain metastases
* Prior radiotherapy within 4 weeks prior to the first day of treatment
* Prior surgery within 3 weeks prior to the first day of treatment
* Prior chemotherapy within 3 weeks prior to the first day of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
maximum tolerated doses of drugs in combination
overall toxicity of drug combination
preliminary antitumor activity of drug combination
impact of pemetrexed on topotecan pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States